CLINICAL TRIAL: NCT05460052
Title: Evaluation of the Effectiveness of a Physical Activity Program on the Severity of Narcolepsy
Acronym: NARCOSPORT
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL21_1430
Record Dates: First submitted 2022-05-23; First posted 2022-07-15 (Actual); Last update posted 2024-01-10 (Actual); Status verified 2024-01

CONDITIONS: Narcolepsy Type 1
Keywords: Narcolepsy; Chronic neurological disorder; Regular physical activity
MeSH Terms: conditions — Narcolepsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Immediate treatment (IT): Patients randomized to the IT group will begin the training sessions 14 days after the inclusion.
  Interventions: Other: Physical activity training program; Other: Personalized training plan.
- Waiting list (WL): Patients randomized to the WL group will receive a weekly phone call for 6 weeks.
  Then, they will benefit the same training program as IT group (56 days after the inclusion).
  Interventions: Other: Physical activity training program; Other: Weekly phone call.; Other: Personalized training plan.

INTERVENTIONS:
Other: Physical activity training program — The physical activity training program will consist of 3 sessions per week for 6 weeks :
  * 1 session will take place in the Sports Medicine Department of the Croix Rousse Hospital
  * 2 sessions will take place remotely. They will be led by an educator in Adapted Physical Activity in live video-conference.
Other: Weekly phone call. — Patients included in the WL group will receive a weekly phone call for 6 weeks (waiting period), before starting the physical activity training program described above.
  Groups: Waiting list (WL)
Other: Personalized training plan. — After the training program, patients of both groups will be given a personalized training plan to be followed for 4 months with regular phone call from the Adapted Physical Activity educator.

SUMMARY:
Narcolepsy Type 1 (NT1) is a rare chronic neurological disorder resulting from the selective loss of hypocretin neurons. Patients with NT1 suffer from excessive daytime sleepiness, disrupted nighttime sleep, and cataplexy (emotionally triggered episodes of muscle atonia). The disease is associated with numerous comorbidities such as obesity, metabolic disorders, anxiety-depressive disorders, and attentional disorders, all of which have a strong impact on quality of life.

DETAILED DESCRIPTION:
Narcolepsy Type 1 (NT1) is a rare chronic neurological disorder resulting from the selective loss of hypocretin neurons. Patients with NT1 suffer from excessive daytime sleepiness, disrupted nighttime sleep, and cataplexy (emotionally triggered episodes of muscle atonia). The disease is associated with numerous comorbidities such as obesity, metabolic disorders, anxiety-depressive disorders, and attentional disorders, all of which have a strong impact on quality of life.

Current management is based on sleep hygiene as well as wake-promoting and anti-cataplectic medications. However, many patients complain of residual sleepiness or cataplexy. In addition, most of the proposed treatments are accompanied by side effects and have little effect on the comorbidities associated with the disease. Therapeutic alternatives are therefore needed in the management of narcolepsy.

Regular Physical Activity (RPA) is recommended by the World Health Organization (WHO) and has been shown to improve anxiety disorders, obesity, metabolic disorders, cognitive functions, sleep and quality of life.

In NT1, patients have fewer opportunities to practice RPA because of daytime sleepiness as well as increased sleep needs. Some studies suggest that cardiorespiratory performances may be lower in NT1 patients than in healthy controls, and that a higher level of physical activity may be associated with lower sleepiness and better metabolic profile in NT1 children. However, no prospective study has evaluated the feasibility of an exercise training program in NT1 or the effect of regular physical activity on disease severity.

The main objective of the study is to evaluate the effect of a physical activity training program of 3 sessions per week for 6 weeks on the severity of narcolepsy in sedentary adults with NT1.

The secondary objectives are to evaluate the feasibility of this program in an adult NT1 population, the effect of the program on comorbidities (obesity, metabolic disorders, anxiety-depressive symptoms, cognitive disorders), medication dosage and quality of life, its tolerance, and the satisfaction of the patients at short- (6 weeks) and long-term (6 months).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Narcolepsy type 1 according to International Classification of Sleep Disorders, 3rd edition (ICSD 3-2014) criteria
* Patients aged 18 to 65 years
* Patients beneficiaries of social security
* Signed consent to participate in the study
* Access to a video conferencing device (smartphone, tablet or computer)

Exclusion Criteria:

* - Patients with a high level of physical activity on the Ricci and Gagnon Questionnaire (score >35) and/or regular physical activity in clubs
* Treatments not stabilized for less than 3 months
* Cognitive disorders incompatible with the understanding and implementation of the program
* Medical contraindication to exercise training
* Patient working night shifts
* Unstable somatic or psychiatric pathology
* Severe untreated obstructive sleep apnea syndrome (apnea/hypopnea index >30/h)
* Pregnancy in progress or breastfeeding
* Persons deprived of liberty by a judicial or administrative decision,
* Persons admitted to a health or social institution for purposes other than research
* Persons of full age who are subject to a legal protection measure or who are unable to express their consent

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with type 1 narcolepsy, sedentary, aged 18 to 65 years. The patients will be recruited from the active file of adult NT1 patients followed in the Sleep Center of the University Hospital of Lyon.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2022-08-26 (Actual); Primary Completion 2023-11-24 (Actual); Study Completion 2023-11-24 (Actual)

PRIMARY OUTCOMES:
Change from baseline Narcolepsy Severity Scale (NSS) Score after training period. | before and after 6 weeks of physical activity program (training period)
  The Narcolepsy Severity Scale is a validated scale exploring the different symptoms of NT1

SECONDARY OUTCOMES:
Narcolepsy Severity Scale (NSS) Score | At 6 months
  The Narcolepsy Severity Scale is a validated scale exploring the different symptoms of NT1
Compliance with the training program. | weekly during the training period (up to 6 weeks)
  It will be expressed as the percentage of sessions completed
Hospital and Anxiety Depression Scale score | At inclusion, at the end of the training program (6 weeks) and at 6 months
Frequency of cataplexy | every week during de training period (6 weeks)
  Items 8and 9 of the NSS are used to assess frequency of cataplexy
Bron/Lyon Attention Stability Test (BLAST) score | Parameters will be measured at inclusion, at the end of the training program (6 weeks)
body mass index | Parameters will be measured at inclusion, at the end of the training program (6 weeks) and at 6 months*
Maximal Oxygen consumption (VO2 max) | Parameters will be measured at inclusion, at the end of the training program (6 weeks)
Fasting blood sugar | Parameters will be measured at inclusion, at the end of the training program (6 weeks) and at 6 months*
Lipid profile | Parameters will be measured at inclusion, at the end of the training program (6 weeks) and at 6 months*
patient satisfaction score | Parameters will be measured at inclusion, at the end of the training program (6 weeks)
sleep efficiency | Parameters will be measured at inclusion, at the end of the training program (6 weeks) and at 6 months*
  Sleep efficiency is defined as the ratio between total sleeping time and time spent in bed
Euroquol 5 dimensions questionnaire score | At inclusion, at the end of the training program (6 weeks) and at 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Laure PETER-DEREX, MD, PhD, Principal Investigator — Hospices Civils de Lyon
Locations (1):
- Service de médecine du sommeil et des maladies respiratoires, Lyon, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ricordeau F, Stauffer E, Putois B, Jaffiol A, Cheylus A, Pouilloux G, Gabriel K, Hoarau E, Bastuji H, Franco P, Herbillon V, Capelle T, Joubert F, Pradat P, Spiegel K, Peter-Derex L. Feasibility and efficacy of exercise training on sleep symptoms and comorbidities in narcolepsy type 1: a prospective interventional study. Sleep. 2026 Jan 13;49(1):zsaf272. doi: 10.1093/sleep/zsaf272. PMID 40928141